CLINICAL TRIAL: NCT06630338
Title: Use of Shear Wave Elastography for Intraoperative Brain and Tumor Stiffness Measurements
Status: Not yet recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 24-003917; NCI-2024-07560 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-003917 (Other: Mayo Clinic in Florida)
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Brain Tumor; Recurrent Brain Tumor; Brain Neoplasm; Recurrent Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients undergo shear wave elastography ultrasound over 10-15 minutes during their standard of care surgery on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study investigates the role of intraoperative shear wave elastography ultrasound (ISWEU) in identifying healthy brain and tumor tissue stiffness differences. This data may be used to guide tumor resection in future patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the feasibility of utilizing ISWEU measurements intraoperatively and in the human brain to measure tissue stiffness.

OUTLINE: This is an observational study.

Patients undergo shear wave elastography ultrasound over 10-15 minutes during their standard of care surgery on study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years old.
* Patients must have planned surgery for resection of a newly diagnosed or recurrent brain tumors.
* Patients with tumors located in the brain cortex or superficial white matter in which introduction of the ultrasound probe is straightforward and does not pose a risk for intraoperative complications.
* Patients must have a Karnofsky performance status ≥ 60%.
* Patient or legally authorized representative (LAR) willing to provide written informed consent.

Exclusion Criteria:

* Patients with deep-seated brain tumors in which introduction of the ultrasound probe poses an increased risk.
* Patients with a history of any brain infections.
* Patients with implanted devices.
* Patients with any other neurological/neurosurgical disease that could affect tissue stiffness.
* Patients with any other structural brain defect that could affect tissue stiffness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults >= 18 years with a brain tumor diagnosis that will undergo brain surgery with tissue resection as standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2033-06-28 (Estimated); Study Completion 2033-06-28 (Estimated)

PRIMARY OUTCOMES:
Feasibility of utilizing Intraoperative Shear Wave Elastography Ultrasound (ISWEU) measurements intraoperatively and in the human brain to measure tissue stiffness. | At baseline
  After intraoperative measurement of brain stiffness using ISWEU, analysis will be conducted after each procedure by determining the tissue stiffness from different areas (tumor core, peritumoral brain zone, and non-cancerous brain tissue) and comparing the tumor stiffness between patients. Reviewers will determine whether ISWEU is feasible to be used as a tool to influence surgical decision.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Quinones-Hinojosa, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials